CLINICAL TRIAL: NCT03488030
Title: Real-world Data of Moderate to Severe Inflammatory Bowel Disease in Argentina: A Non-interventional, Multicenter Study to Evaluate Disease Control, Treatment Patterns, Burden of Disease and Quality of Life
Brief Title: A Study to Evaluate Disease Control, Treatment Patterns, Burden of Disease and Quality of Life in Participants With Moderate to Severe Inflammatory Bowel Disease (IBD)
Acronym: RISE AR
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: IBD-5004; U1111-1207-4110 (Other: WHO)
Record Dates: First submitted 2018-03-27; First posted 2018-04-04 (Actual); Results first posted 2020-06-12 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Disease
Keywords: Drug therapy
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: Participants diagnosed with moderate to severe UC or CD from the 7 participating sites will be observed on Day 1 for cross-sectional evaluation of disease activity, treatment patterns, burden of disease and quality of life along with retrospective data collection for previous 3 years from the date of UC or CD diagnosis until Day 1 to assess the IBD treatments, medical history and comorbidities, treatment patterns and use of health resources.

SUMMARY:
The purpose of this study is to evaluate the percentage of moderate to severe IBD participants with active disease at Day 1.

DETAILED DESCRIPTION:
This is a retrospective, cross-sectional, and non-interventional study of participants with IBD. The study will have a cross-sectional evaluation on Day 1 to provide the real-world data of disease activity, treatment patterns, burden of disease and quality of life in participants with moderate to severe CD or UC.

The study will involve an additional retrospective review of medical charts of participants of previous 3 years to describe the IBD treatments and use of other healthcare resources related with management of IBD.

The study will enroll approximately 246 participants. All participants will be enrolled in one observational cohort.

This multi-center trial will be conducted in Argentina. The overall time for data collection in the study will be approximately 3 years before the start of the study (Day 1).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of moderate to severe CD or UC for at least 6 months prior to Day 1 appointment based on clinical or endoscopic or image criteria.

Exclusion Criteria:

1. Indeterminate or not classified colitis.
2. Presenting mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with moderate to severe CD or UC will be observed.
Sampling Method: Non-Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (7):
- Argentina (7):
  - Centro de Educacion Medica e Investigaciones Clinicas Norberto Quirno (CEMIC), CABA, Buenos Aires
  - Hospital Britanico de Buenos Aires, CABA, Buenos Aires
  - Hospital de Gastroenterologia Dr. Carlos Bonorino Udaondo, CABA, Buenos Aires
  - Sanatorio Mater Dei, CABA, Buenos Aires
  - Hospital San Martin, La Plata, Buenos Aires
  - Hospital Provincial del Centenario, Rosario, Santa Fe Province
  - Hospital Privado de Cordoba, Córdoba

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Result] Olivera PA, Balderramo D, Lasa JS, Zubiaurre I, Correa G, Lubrano P, Ruffinengo O, Yantorno M, Rausch A, Pinero G, Bolomo A, Amigo C, El-Hakeh J, Leonardi DB, Brion L, Sambuelli A. Real-world clinical characteristics and therapeutic strategies in patients with moderate-to-severe inflammatory bowel disease in Argentina: Data from the RISE-AR study. Gastroenterol Hepatol. 2025 Oct;48(8):502287. doi: 10.1016/j.gastrohep.2024.502287. Epub 2024 Nov 15. English, Spanish. PMID 39549817
- [Result] P426 Health-Related Quality of Life and Work Productivity in patients with moderate-to-severe Inflammatory Bowel Disease in Argentina: Data from the RISE AR study. G J Correa, M Yantorno, P Olivera Sendra, J S Lasa, P Lubrano, D C Balderramo, I Zubiaurre, O Ruffinengo, L Brion, D B Leonardi, J El-Hakeh, P N Guimaraens, A Sambuelli. Journal of Crohn's and Colitis, Volume 15, Issue Supplement_1, May 2021, Pages S430-S431, https://doi.org/10.1093/ecco-jcc/jjab076.550

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 7 investigative sites in Argentina from 12 December 2018 to 31 May 2019.
Pre-assignment Details: Participants diagnosed with moderate to severe Inflammatory Bowel Disease (IBD)- Crohn's disease (CD) or ulcerative colitis (UC) were observed on Day 1 with retrospective data collection for previous 3 years.
Groups:
- Crohn's Disease: Participants diagnosed with moderate to severe CD for at least 6 months prior to Day 1 appointment from the 7 participating sites were observed on Day 1 for cross-sectional evaluation of disease activity, treatment patterns, burden of disease and quality of life along with retrospective data collection for previous 3 years from the date of CD diagnosis until Day 1 to assess the IBD treatments, medical history and comorbidities, treatment patterns and use of health resources.
- Ulcerative Colitis: Participants diagnosed with moderate to severe UC for at least 6 months prior to Day 1 appointment from the 7 participating sites were observed on Day 1 for cross-sectional evaluation of disease activity, treatment patterns, burden of disease and quality of life along with retrospective data collection for previous 3 years from the date of UC diagnosis until Day 1 to assess the IBD treatments, medical history and comorbidities, treatment patterns and use of health resources.
Period: Overall Study
Arm/Group | Crohn's Disease | Ulcerative Colitis
Started | 101 | 145
Completed (Participants with moderate to severe IBD at Day 1.) | 101 | 145
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis dataset by IBD included all participants fulfilling selection criteria, who provided the written informed consent, without major study protocol deviations and who had completed the Day 1 assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Crohn's Disease | Ulcerative Colitis | Total
Number analyzed (Participants) | 101 | 145 | 246
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.92 (14.50) | 45.61 (15.83) | 44.51 (15.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 79 | 130
  Male | 50 | 66 | 116
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 101 | 145 | 246
Professional Situation [Count of Participants; unit: Participants] — Participants were stratified by the following categories: employed, unemployed, student, retired, other, and unknown.
  Participants
    Employed | 66 | 88 | 154
    Unemployed | 12 | 17 | 29
    Student | 4 | 6 | 10
    Retired | 11 | 23 | 34
    Other | 7 | 11 | 18
    Unknown | 1 | 0 | 1
Educational Level [Count of Participants; unit: Participants] — Participants were stratified by the following categories: not literate, primary school, primary school not completed, secondary school, secondary school not completed, higher education, higher education not completed, post-graduate or Master of Business Administration (MBA), and unknown.
  Participants
    Not literate | 0 | 0 | 0
    Primary school | 5 | 6 | 11
    Primary school not completed | 0 | 4 | 4
    Secondary school | 25 | 33 | 58
    Secondary school not completed | 8 | 17 | 25
    Higher education | 40 | 59 | 99
    Higher education not completed | 18 | 17 | 35
    Post-graduate or MBA | 4 | 8 | 12
    Unknown | 1 | 1 | 2
Participant's Income [Count of Participants; unit: Participants] — Participants were stratified by the following categories: no income, from 30 dollar to 3.700 dollar, from 3.700 dollar to 6.000 dollar, from 6.000 dollar to 7.100 dollar, from 7.100 dollar to 8.500 dollar, from 8.500 dollar to 11.000 dollar, from 11.000 dollar to 13.800 dollar, from 13.800 dollar to 16.000 dollar, from 16.000 dollar to 20.000 dollar, from 20.000 dollar to 29.000 dollar, from 29.000 dollar to 800.000 dollar and unknown.
  Participants
    No income | 15 | 22 | 37
    From 30 dollar to 3.700 dollar | 1 | 0 | 1
    From 3.700 dollar to 6.000 dollar | 0 | 2 | 2
    From 6.000 dollar to 7.100 dollar | 0 | 0 | 0
    From 7.100 dollar to 8.500 dollar | 3 | 1 | 4
    From 8.500 dollar to 11.000 dollar | 7 | 10 | 17
    From 11.000 dollar to 13.800 dollar | 1 | 3 | 4
    From 13.800 dollar to 16.000 dollar | 4 | 5 | 9
    From 16.000 dollar to 20.000 dollar | 4 | 9 | 13
    From 20.000 dollar to 29.000 dollar | 6 | 12 | 18
    From 29.000 dollar to 800.000 dollar | 26 | 43 | 69
    Unknown | 34 | 38 | 72
Smoking Status [Count of Participants; unit: Participants] — Participants were stratified by the following categories: never smoked or smoked less than 100 cigarettes, former smoker and current smoker.
  Participants
    Never smoked OR smoked less than 100 cigarettes | 57 | 84 | 141
    Former smoker | 31 | 53 | 84
    Current smoker | 13 | 8 | 21
Family History of IBD [Count of Participants; unit: Participants] — Participants were stratified by the following categories: with IBD history, without IBD history, and unknown.
  Participants
    With IBD history | 12 | 8 | 20
    Without IBD history | 88 | 135 | 223
    Unknown | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Crohn's Disease: Percentage of Participants With Active CD at Day 1
Description: Percentage of participants with active CD were observed, where active CD was defined as Harvey Bradshaw index (HBI) greater than or equal to (>=) 8 or Crohn's disease active index (CDAI) >= 220 points. CDAI assessed CD based on clinical signs and symptoms such as number of liquid stools, intensity of abdominal pain, general wellbeing, presence of comorbid conditions, use of antidiarrheal, physical examination and laboratory findings. Total score ranged from 0 to 600 points. Higher score indicated more severe disease. HBI consisted of 5 clinical parameters: general well-being, abdominal pain, number of liquid stools per day, abdominal mass, and complications. Total score was sum of individual parameters. Score ranges from a minimum score of 0 to no pre-specified maximum score as it depends on number of liquid stools, where higher scores indicated more severe disease.
Time Frame: Day 1
Population: Analysis dataset for disease activity included all participants who fulfilled selection criteria, provided the written informed consent, were without major study protocol deviations, had completed the Day 1 assessment, and who had no ostomy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Crohn's Disease
Number analyzed (Participants) | 97
percentage of participants | 9.3 [4.3 to 16.9]

2. Primary Outcome: Ulcerative Colitis: Percentage of Participants With Active UC at Day 1
Description: Percentage of participants with active disease UC disease were observed, where UC was defined as 9-point Partial Mayo Score (pMayo score) >=5. The Mayo score was composed of four categories (bleeding, stool frequency, physician assessment, and endoscopic appearance) rated from 0 to 3 that are summed to give a total score that ranges from 0 to 12. The pMayo score was previously compared with the full Mayo score and categorized participants as being in remission (score of 0 to 2), having mild disease (pMayo of 3 or 4) or moderate to severe disease (pMayo of >=5).
Time Frame: Day 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ulcerative Colitis
Number analyzed (Participants) | 143
percentage of participants | 7.7 [3.9 to 13.3]

3. Secondary Outcome: Number of Participants With Moderate to Severe CD or UC Stratified by Steroid Behavior
Time Frame: Day 1
Population: Analysis dataset by IBD included all participants who fulfilled selection criteria, provided the written informed consent, were without major protocol deviations, and who had completed the Day 1 assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Crohn's Disease | Ulcerative Colitis
Number analyzed (Participants) | 101 | 145
Participants
  Steroid-dependent | 28 | 71
  Steroid-refractory disease | 16 | 12
  Not applicable (who did not use previously) | 5 | 7
  Steroid-responsive disease | 52 | 54
  Unknown | 0 | 1

4. Secondary Outcome: Number of Participants With Moderate to Severe CD or UC Stratified by Anthropometric Information
Description: Anthropometric information included height, weight and body mass index (BMI). BMI ranges: underweight (BMI less than [<] 18.50 kilogram per square meter (kg/m^2), normal range (BMI between 18.50 and 24.99 kg/m^2), overweight (BMI between 25.00 and 29.99 kg/m^2), obese (BMI >=30.00 kg/m^2).
Time Frame: Day 1
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Crohn's Disease | Ulcerative Colitis
Number analyzed (Participants) | 101 | 145
Participants
  Height (cm) | NA — Data was not collected according to the pre-defined categories. | NA — Data was not collected according to the pre-defined categories.
  Weight (kg) | NA — Data was not collected according to the pre-defined categories. | NA — Data was not collected according to the pre-defined categories.
  BMI, underweight | 3 | 8
  BMI, normal range | 54 | 55
  BMI, overweight | 33 | 55
  BMI, obese | 11 | 27

5. Secondary Outcome: Number of Participants With Moderate to Severe CD or UC Based on Medical History, Comorbidities or Extra Intestinal Manifestation (EIM)
Description: Medical history was defined as an EIM or non-EIM according to the investigator's judgement.
Time Frame: Day 1
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Crohn's Disease | Ulcerative Colitis
Number analyzed (Participants) | 101 | 145
Participants
  With medical history, comorbidity or EIM | 49 | 74
  Without medical history, comorbidity or EIM | 52 | 71

6. Secondary Outcome: Crohn's Disease: Number of Participants With Moderate to Severe CD Stratified by Clinical Characterization
Description: The Montreal classification index for CD was used to classify the extent of the disease activity. It consisted of two parameters: location and behavior of the disease activity. There were four different disease locations presented: Location 1 (L1) is ileum, Location 2 (L2) is colonic disease, Location 3 (L3) is ileocolon and Location 4 (L4) is isolated upper gastrointestinal (GI) tract disease. The first three categories (L1-L3) was combined with L4 where disease sites coexisted. There were 4 different categories for the behavior of the disease activity: Behavior 1 (B1) was non stenosing or non penetrating; Behavior 2 (B2) was stenosing; Behavior 3 (B3) was penetrating and p as perianal disease (p). The first 3 categories (B1 to B3) could be added with p to indicate coexisting perianal disease. Perianal disease (p) was defined as the presence of perianal abscesses or fistulae.
Time Frame: Day 1
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Crohn's Disease
Number analyzed (Participants) | 101
Participants
  Location, L1 | 9
  Location, L1+L4 | 2
  Location, L2 | 52
  Location, L2+L4 | 0
  Location, L3 | 33
  Location, L3+L4 | 4
  Location, L4 | 1
  Behavior, B1 | 35
  Behavior, B1+P | 14
  Behavior, B2 | 23
  Behavior, B2+P | 15
  Behavior, B3 | 9
  Behavior, B3+P | 5
  Behavior, P | 0

7. Secondary Outcome: Ulcerative Colitis: Number of Participants With Moderate to Severe CD Stratified by Clinical Characterization
Description: Montreal classification index for UC was used to classify the extent and severity of the disease activity. There were three subgroups of UC defined by extent of inflammation: Extent 1 (E1) =Ulcerative distal UC proctitis and proctosigmoiditis, Extent 2 (E2) =Left-sided mucosa inflammation extending up to splenic flexure and Extent 3 (E3) =Pancolitis mucosa inflammation up to proximal transverse colon and beyond. Severity of UC as S0=Clinical remission (asymptomatic),S1 =Mild UC (passage of four or fewer stools/day [with or without blood],absence of any systemic illness, and normal inflammatory markers),S2 =Moderate UC (passage of more than four stools per day but with minimal signs of systemic toxicity),S3 =Severe UC (passage of at least 6 bloody stools daily, pulse rate of at least 90 beats per minute, temperature of at least 37.5 degree Celsius, hemoglobin of <10.5 gram per 100 milliliter (g/100mL), and erythrocyte sedimentation rate (ESR) of at least 30 millimeter per hour (mm/h).
Time Frame: Day 1
Population: Analysis dataset by IBD included all participants who fulfilled selection criteria, provided the written informed consent, were without major protocol deviations, and who had completed the Day 1 assessment. Here "overall number of participants analyzed" are participants who were available for this outcome measure assessment at given time period.
Measure: Count of Participants; unit: Participants
Arm/Group | Ulcerative Colitis
Number analyzed (Participants) | 143
Participants
  Extent Inflammation, E1-Distal: Proctitis | 13
  Extent Inflammation, E1-Distal: Proctosigmoiditis | 4
  Extent of Inflammation, E2 | 60
  Extent of Inflammation, E3 | 66
  Severity, S0 | 66
  Severity, S1 | 33
  Severity, S2 | 30
  Severity, S3 | 14

8. Secondary Outcome: Number of Participants With Moderate to Severe CD or UC Who Used Various Types of Therapies for IBD in Previous 3 Years
Description: Various types of therapies for IBD included salicylic derivatives, corticosteroids, immunosuppressors, biologic therapy, antibiotics, nutrition support and others. One participant could use more than one therapy.
Time Frame: Within previous 3 years including Day 1
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Crohn's Disease | Ulcerative Colitis
Number analyzed (Participants) | 101 | 145
Participants
  Salicylic derivatives | 63 | 142
  Corticosteroids | 56 | 101
  Immunosuppressors | 66 | 85
  Biologic therapy | 80 | 49
  Antibiotics | 14 | 13
  Nutrition support | 0 | 0
  Other | 9 | 25

9. Secondary Outcome: Duration of IBD Treatment During Previous 3 Years
Description: Time between the beginning of IBD treatment until the end of treatment. For participants with ongoing IBD treatment at Day 1, stop date was considered as Day 1 date visit. Various types of therapies for IBD included salicylic derivates, corticosteroids, immunosuppressors, biologic therapy, antibiotics, nutrition support and others. One participant could use more than one therapy.
Time Frame: Within previous 3 years including Day 1
Population: Analysis dataset by IBD included all participants who fulfilled selection criteria, provided the written informed consent, were without major protocol deviations, and who had completed the Day 1 assessment. Participants available for this outcome measure at given time period were included for assessment.
Measure: Median (Full Range); unit: months
Arm/Group | Crohn's Disease | Ulcerative Colitis
Number analyzed (Participants) | 101 | 145
months
  Salicylic derivates treatment: number analyzed (Participants) | 63 | 141
  Salicylic derivates treatment | 35.90 [0.52 to 35.97] | 33.11 [0.03 to 35.97]
  Corticosteroids treatment: number analyzed (Participants) | 55 | 98
  Corticosteroids treatment | 3.74 [0.03 to 35.97] | 3.96 [0.03 to 35.97]
  Immunosuppressors treatment: number analyzed (Participants) | 66 | 84
  Immunosuppressors treatment | 21.13 [0.03 to 35.97] | 19.54 [0.03 to 35.97]
  Biologic therapy treatment: number analyzed (Participants) | 80 | 49
  Biologic therapy treatment | 29.26 [0.03 to 35.97] | 17.97 [0.03 to 35.97]
  Antibiotics treatment: number analyzed (Participants) | 14 | 12
  Antibiotics treatment | 1.33 [0.26 to 35.97] | 0.59 [0.07 to 1.28]

10. Secondary Outcome: Number of Participants With Moderate to Severe CD or UC Treated With Biologic Therapy During Previous 3 Years
Description: Biologic therapies included infliximab, adalimumab, vedolizumab, certolizumab, golimumab, and ustekimumab. For participants with ongoing biologic therapy at Day 1, stop date was considered as Day 1 date visit.
Time Frame: Within previous 3 years including Day 1
Population: Analysis dataset by IBD included all participants who fulfilled selection criteria, provided written informed consent, were without major protocol deviations, and who had completed Day 1 assessment. Here "overall number of participants analyzed" are participants who had biologic therapies, and who were available for assessment at given time period.
Measure: Count of Participants; unit: Participants
Arm/Group | Crohn's Disease | Ulcerative Colitis
Number analyzed (Participants) | 71 | 43
Participants
  Infliximab | 17 | 23
  Adalimumab | 51 | 18
  Vedolizumab | 2 | 1
  Certolizumab | 1 | 0
  Golimumab | 0 | 1
  Ustekimumab | 0 | 0

11. Secondary Outcome: Number of Participants With Moderate to Severe CD or UC Who Have Not Responded Previously to Biologic Therapies With Reasons
Time Frame: Within previous 3 years including Day 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Crohn's Disease | Ulcerative Colitis
Number analyzed (Participants) | 97 | 143
Participants
  Adverse reaction | 4 | 0
  Pregnancy | 1 | 2
  Surgery | 4 | 0
  Poor effectiveness | 16 | 8
  Remission | 2 | 0
  Patient decision | 0 | 3
  Patient poor adherence | 1 | 0
  Patient access to treatment | 1 | 1
  Other | 0 | 1
  End of treatment as expected | 0 | 1

12. Secondary Outcome: Number of Participants With Moderate to Severe CD or UC Who Had IBD Treatment Initiation on Day 1
Time Frame: Day 1
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Crohn's Disease | Ulcerative Colitis
Number analyzed (Participants) | 101 | 145
Participants | 11 | 20

13. Secondary Outcome: Number of Participants With Moderate to Severe and No or Mild Activity of CD or UC Stratified by Socio-demographic Variables
Description: Participants were stratified based on gender, professional status, educational level and income.
Time Frame: Day 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Crohn's Disease (Moderate to Severe): Participants diagnosed with moderate to severe CD (HBI score >=8 points and CDAI score >=220 points) for at least 6 months prior to Day 1 appointment from the 7 participating sites were observed on Day 1 for cross-sectional evaluation of disease activity, treatment patterns, burden of disease and quality of life along with retrospective data collection for previous 3 years from the date of CD diagnosis until Day 1 to assess the IBD treatments, medical history and comorbidities, treatment patterns and use of health resources.
- Crohn's Disease (no or Mild): Participants diagnosed with no or mild CD (HBI score <8 points and CDAI score < 220 points) from the 7 participating sites will be observed on Day 1 for cross-sectional evaluation of disease activity, treatment patterns, burden of disease and quality of life along with retrospective data collection for previous 3 years from the date of CD diagnosis until Day 1 to assess the IBD treatments, medical history and comorbidities, treatment patterns and use of health resources.
- Ulcerative Colitis (Moderate to Severe): Participants diagnosed with moderate to severe UC (9-point pMayo score >=5) for at least 6 months prior to Day 1 appointment from the 7 participating sites were observed on Day 1 for cross-sectional evaluation of disease activity, treatment patterns, burden of disease and quality of life along with retrospective data collection for previous 3 years from the date of UC diagnosis until Day 1 to assess the IBD treatments, medical history and comorbidities, treatment patterns and use of health resources.
- Ulcerative Colitis (no or Mild): Participants diagnosed with no or mild UC (9-point pMayo score <5) from the 7 participating sites will be observed on Day 1 for cross-sectional evaluation of disease activity, treatment patterns, burden of disease and quality of life along with retrospective data collection for previous 3 years from the date of UC diagnosis until Day 1 to assess the IBD treatments, medical history and comorbidities, treatment patterns and use of health resources.
Arm/Group | Crohn's Disease (Moderate to Severe) | Crohn's Disease (no or Mild) | Ulcerative Colitis (Moderate to Severe) | Ulcerative Colitis (no or Mild)
Number analyzed (Participants) | 9 | 88 | 11 | 132
Participants
  Gender, male | 3 | 44 | 3 | 61
  Gender, female | 6 | 44 | 8 | 71
  Professional status, employed | 5 | 58 | 6 | 81
  Professional status, unemployed | 1 | 11 | 2 | 15
  Professional status, student | 0 | 4 | 0 | 6
  Professional status, retired | 2 | 9 | 1 | 21
  Professional status, other | 1 | 5 | 2 | 9
  Professional status, unknown | 0 | 1 | 0 | 0
  Educational level, not literate | 0 | 0 | 0 | 0
  Educational level, primary school | 0 | 4 | 0 | 5
  Educational level, primary school not completed | 0 | 0 | 1 | 3
  Educational level, secondary school | 4 | 20 | 2 | 31
  Educational level, secondary school not completed | 1 | 6 | 1 | 16
  Educational level, higher school | 2 | 38 | 6 | 52
  Educational level, higher school not completed | 1 | 16 | 0 | 17
  Educational level, Post-graduate/MBA | 1 | 3 | 1 | 7
  Educational level, missing values | 0 | 1 | 0 | 1
  Income, no income | 1 | 14 | 3 | 19
  Income, from 30 dollar to 3.700 dollar | 1 | 0 | 0 | 0
  Income, from 3.700 dollar to 6.000 dollar | 0 | 0 | 0 | 2
  Income, from 6.000 dollar to 7.100 dollar | 0 | 0 | 0 | 0
  Income, from 7.100 dollar to 8.500 dollar | 1 | 2 | 0 | 1
  Income, from 8.500 dollar to 11.000 dollar | 2 | 5 | 2 | 7
  Income, from 11.000 dollar to 13.800 dollar | 0 | 0 | 0 | 3
  Income, from 13.800 dollar to 16.000 dollar | 0 | 3 | 0 | 5
  Income, from 16.000 dollar to 20.000 dollar | 0 | 4 | 1 | 8
  Income, from 20.000 dollar to 29.000 dollar | 0 | 6 | 1 | 11
  Income, from 29.000 dollar to 800.000 dollar | 1 | 23 | 2 | 40
  Income, from unknown values | 3 | 31 | 2 | 36

14. Secondary Outcome: Quality of Life Assessed by European Quality of Life 5-dimension (EQ-5D) Health States Visual Analogue Scale (VAS) Score at Day 1
Description: EQ-5D considered five attributes of quality of life evaluation, that is, mobility, self-care, usual activity, pain/discomfort, and anxiety/depression. Each dimension had five possible levels: 1 (no problems); 2 (slight problems); 3 (moderate problems); 4 (severe problems), and; 5 (extreme problems). EQ-5D also included an additional visual analogic scale (EQ-VAS), which ranged from 0 to 100, where 0 indicated worst imaginable health state and 100 was best imaginable health state.
Time Frame: Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crohn's Disease | Ulcerative Colitis
Number analyzed (Participants) | 101 | 145
score on a scale | 74.82 (17.37) | 75.74 (16.40)

15. Secondary Outcome: Quality of Life as Assessed by 36-item Short Form Health Survey (SF-36) Component Score at Day 1
Description: The SF-36 evaluated 8 health dimensions: physical functioning, bodily pain, role physical (limitations due to physical problems), role emotional (limitations due to personal or emotional problems), mental health, social functioning, vitality, and general health perceptions. Based on these 4 scales (physical functioning, role-physical, bodily pain, general health), the physical component summary (PCS) score was generated which ranged between 0 and 100, with higher scores indicating a better quality of life. Based on these 4 scales (vitality, social functioning, role-emotional, and mental health), the mental component summary (MCS) score was generated which ranged between 0 and 100, with higher scores indicating a better quality of life.
Time Frame: Day 1
Population: Analysis dataset by IBD included all participants who fulfilled selection criteria, provided the written informed consent, were without major protocol deviations, and who had completed the Day 1 assessment. Participants available for this outcome measure at given time period were included for the assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crohn's Disease | Ulcerative Colitis
Number analyzed (Participants) | 101 | 145
score on a scale
  MCS score: number analyzed (Participants) | 101 | 143
  MCS score | 43.61 (11.27) | 45.85 (10.09)
  PCS score: number analyzed (Participants) | 101 | 143
  PCS score | 50.47 (7.95) | 50.37 (7.06)

16. Secondary Outcome: Inflammatory Bowel Disease Questionnaire (IBDQ) Total Score at Day 1
Description: The IBDQ was a 32-item questionnaire that measured 4 dimensions: bowel function, emotional status, systemic symptoms, and social function. Within dimensions, each question presented seven possible answers/points. Each domain score was the sum of 8 responses each ranging from 1 to 7, where 1 indicated worst function and 7 the best. The sub-score ranged from 8 to 56 and thus the total score ranged from 32 to 224, where higher score indicating better quality of life.
Time Frame: Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crohn's Disease | Ulcerative Colitis
Number analyzed (Participants) | 101 | 145
score on a scale | 22.07 (4.64) | 22.38 (4.30)

17. Secondary Outcome: Inflammatory Bowel Disease Questionnaire (IBDQ) Domain Score at Day 1
Description: IBDQ was a 32-item questionnaire that measured 4 dimensions: bowel systems, emotional health, systemic systems, and social function. Within dimensions, each question presented seven possible answers/points. Each domain score was the average of 8 responses each ranging from 1 to 7, where 1 indicated worst function and 7 the best function.
Time Frame: Day 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Crohn's Disease | Ulcerative Colitis
Number analyzed (Participants) | 101 | 145
score on scale
  Bowel systems: number analyzed (Participants) | 97 | 141
  Bowel systems | 5.64 (1.18) | 5.73 (1.10)
  Emotional health: number analyzed (Participants) | 97 | 141
  Emotional health | 5.21 (1.40) | 5.38 (1.25)
  Systemic systems: number analyzed (Participants) | 97 | 142
  Systemic systems | 5.15 (1.16) | 5.15 (1.21)
  Social function: number analyzed (Participants) | 94 | 139
  Social function | 6.02 (1.40) | 5.96 (1.32)

18. Secondary Outcome: Mean of Percentage of Total Work Productivity Impairment (TWPI) Due to CD or UC as Assessed by Work Productivity and Activity Impairment Questionnaire (WPAI)
Description: WPAI assessed impact of IBD on work productivity and daily activities in past 7 days. WPAI questions were: if currently employed, 2) hours (hrs) missed due to disease, 3) hrs missed other reasons, 4) hrs actually worked, 5) degree disease affected productivity while working, 6) degree disease affected regular activities. WPAI generates 4 component scores: percentage (%) of work time missed (absenteeism), % of impairment while working (presenteeism), % of overall work impairment (absenteeism and presenteeism combined), and % of activity impairment. TWPI was calculated based on 3 items: (Q2) number of hrs missed from work due to health problems in the past 7 days; (Q4) number of actual work hrs in past 7 days; and (Q5) to what degree did disease impair productivity while working in past 7 days. Data was calculated by: Q2/(Q2+Q4)+([1-(Q2/[Q2+Q4])*(Q5/10])*100 (converted to %). Data is presented as impairment percentage, with higher numbers indicating greater impairment/less productivity.
Time Frame: Day 1
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percentage of TWPI
Arm/Group | Crohn's Disease | Ulcerative Colitis
Number analyzed (Participants) | 58 | 81
Percentage of TWPI | 98.83 (3.27) | 98.79 (4.06)

19. Secondary Outcome: Mean of Percentage of Work Time Missed Due to CD or UC as Assessed by WPAI at Day 1
Description: WPAI assessed impact of IBD on work productivity and daily activities in past 7 days. WPAI questions were: if currently employed, 2) hours missed due to disease, 3) hours missed other reasons, 4) hours actually worked, 5) degree disease affected productivity while working, 6) degree disease affected regular activities. WPAI generates 4 component scores: percentage of work time missed (absenteeism), percentage of impairment while working (presenteeism), percentage of overall work impairment (absenteeism and presenteeism combined), and percentage of activity impairment. Work time missed was calculated based on 2 items: (Q2) number of hours missed from work due to health problems in the past 7 days; and (Q4) number of actual work hours in past 7 days. Data was calculated by following formula:Q2/(Q2+Q4)*100 (converted to %), where higher numbers indicated greater impairment and less productivity.
Time Frame: Day 1
Population: Analysis dataset by IBD included all participants who fulfilled selection criteria, provided the written informed consent, were without major protocol deviations, and who had completed the Day 1 assessment. Here "overall number of participants analyzed" are participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of work time missed
Arm/Group | Crohn's Disease | Ulcerative Colitis
Number analyzed (Participants) | 62 | 85
percentage of work time missed | 9.65 (25.38) | 7.81 (22.45)

20. Secondary Outcome: Mean of Percentage of Impairment While Working Due to CD or UC as Assessed by WPAI at Day 1
Description: WPAI assessed impact of IBD on work productivity and daily activities in past 7 days. WPAI questions were: if currently employed, 2) hours missed due to disease, 3) hours missed other reasons, 4) hours actually worked, 5) degree disease affected productivity while working, 6) degree disease affected regular activities. WPAI generates 4 component scores: percentage of work time missed (absenteeism), percentage of impairment while working (presenteeism), percentage of overall work impairment (absenteeism and presenteeism combined), and percentage of activity impairment. Percentage of impairment while working was calculated based on 1 item: (Q5) to what degree did disease impair productivity while working in past 7 days. The item was measured on a scale from 0 (no effect) to 10 (completely prevented from doing regular activities/ working). Data was calculated by following formula: Q5/10*100 (converted to percent), where higher numbers indicated greater impairment and less productivity.
Time Frame: Day 1
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: percentage of impairment while working
Arm/Group | Crohn's Disease | Ulcerative Colitis
Number analyzed (Participants) | 58 | 82
percentage of impairment while working | 10.86 (19.04) | 11.95 (18.08)

21. Secondary Outcome: Mean of Percentage of Total Activity Impairment Due to CD or UC as Assessed by WPAI at Day 1
Description: WPAI assessed impact of IBD on work productivity and daily activities in past 7 days. WPAI questions were: if currently employed, 2) hours (hrs) missed due to disease, 3) hrs missed other reasons, 4) hrs actually worked, 5) degree disease affected productivity while working, 6) degree disease affected regular activities. WPAI generates 4 component scores: percentage (%) of work time missed (absenteeism), % of impairment while working (presenteeism), % of overall work impairment (absenteeism and presenteeism combined), and % of activity impairment. % of total activity impairment was calculated based on: (Q6) in past 7 days, how much did your health problems affect your ability to do your regular daily activities, other than work at a job. Item was measured on scale from 0 (no effect) to 10 (completely prevented from doing regular activities/ working). Data was calculated by: Q6/10*100 (converted to percent), where higher numbers indicated greater impairment and less productivity.
Time Frame: Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of activity impairment
Arm/Group | Crohn's Disease | Ulcerative Colitis
Number analyzed (Participants) | 101 | 145
percentage of activity impairment | 21.49 (28.09) | 22.62 (27.81)

22. Secondary Outcome: Percentage of Participants Who Quit Job Due to IBD and Have Not Been Able to Return to Work
Time Frame: Day 1
Population: Due to change in planned analysis, data was not collected and analyzed. Percentage of participants who quit job due to IBD and have not been able to return to work was not calculated since this variable was not captured in case report form.
Arm/Group | Crohn's Disease | Ulcerative Colitis
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Number of Participants With Moderate to Severe CD or UC Who Used Healthcare Resources Over the Previous 3 Years
Description: Healthcare resources included drug therapies, imaging and laboratory testing, surgeries, hospitalizations and consultations.
Time Frame: Within previous 3 years including Day 1
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Crohn's Disease | Ulcerative Colitis
Number analyzed (Participants) | 101 | 145
participants
  Previous imaging and laboratory | 100 | 141
  Previous surgeries | 18 | 2
  Previous hospitalization | 34 | 31
  Previous consultation | 98 | 138

ADVERSE EVENTS:
Time Frame: Not applicable, as safety data was not planned to be collected during the study
Description: Safety data was not planned to be collected in this observational retrospective study.
Arm/Group | Crohn's Disease | Ulcerative Colitis
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-01-24): https://cdn.clinicaltrials.gov/large-docs/30/NCT03488030/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-28): https://cdn.clinicaltrials.gov/large-docs/30/NCT03488030/SAP_001.pdf